CLINICAL TRIAL: NCT00970814
Title: A Phase 2, Double Blind, Placebo Controlled Trial to Assess the Efficacy Of Levetiracetam Extended Release in Very Heavy Drinkers
Brief Title: Levetiracetam XR in Very Heavy Drinkers
Acronym: NCIG 002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAA_DTRR-2009-LITTEN-02
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Alcoholism
Keywords: Alcoholism; Alcohol Drinking; Alcoholic Intoxication; Alcohol Abuse
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alcoholic Intoxication | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levetiracetam XR (Active Comparator): Group received Levetiracetam
  Interventions: Behavioral: BBCET; Drug: Levetiracetam XR
- Sugar Pill (Placebo Comparator): Placebo
  Interventions: Behavioral: BBCET; Drug: Sugar Pill

INTERVENTIONS:
Behavioral: BBCET — 11 BBCET sessions
  Arms: Levetiracetam XR
Behavioral: BBCET — 11 BBCET Sessions
  Arms: Sugar Pill
Drug: Levetiracetam XR — 500mg - 2000mg Once per day 16 weeks
  Arms: Levetiracetam XR
Drug: Sugar Pill — 500mg - 2000mg Once per day 16 weeks
  Arms: Sugar Pill

SUMMARY:
The primary objectives of this study are to assess the efficacy of levetiracetam XR in increasing the percentage of subjects with no heavy drinking days and in reducing the weekly percentage of heavy drinking days in subjects with alcohol dependence confirmed by DSM-IV criteria and who frequently consume 10 or more drinks per drinking day for men and 8 or more drinks per drinking day for women (designated as "very heavy" drinkers).

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be at least 18 years of age.
2. The subject must have a DSM-IV diagnosis of current alcohol dependence.
3. The subject must be seeking treatment for alcohol dependence and desires a reduction or cessation of drinking.
4. The subject must be able to verbalize understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
5. If the subject is female and of child bearing potential, she must agree to use at least one of the following methods of birth control, or she must be surgically sterile or postmenopausal:

   * oral contraceptives
   * contraceptive sponge
   * patch
   * barrier (diaphragm or condom)
   * intrauterine contraceptive system
   * levonorgestrel implant
   * medroxyprogesterone acetate contraceptive injection
   * complete abstinence from sexual intercourse, and/or
   * hormonal vaginal contraceptive ring.
6. The subject must be able to take oral medication, willing to adhere to the medication regimen, and willing to return for regular visits.
7. The subject must complete all psychological assessments required at screening and baseline.
8. The subject must provide evidence of stable residence in the last 2 months prior to randomization, have reasonable transportation arrangements to the study site, and have no plans to move within the next 3 months or unresolved legal problems. Subjects must provide contact information of someone, such as a family member, spouse, or significant other, who may be able to contact the subject in case of a missed clinic appointment.
9. The subject must have a breath alcohol concentration (BAC) equal to 0.000 when s/he signed the informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Z Litten, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA); Margaret M Mattson, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA); Joanne E Fertig, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (5):
- United States (5):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Dartmouth Medical School, Lebanon, New Hampshire
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Result] Fertig JB, Ryan ML, Falk DE, Litten RZ, Mattson ME, Ransom J, Rickman WJ, Scott C, Ciraulo D, Green AI, Tiouririne NA, Johnson B, Pettinati H, Strain EC, Devine E, Brunette MF, Kampman K, A Tompkins D, Stout R; NCIG 002 Study Group. A double-blind, placebo-controlled trial assessing the efficacy of levetiracetam extended-release in very heavy drinking alcohol-dependent patients. Alcohol Clin Exp Res. 2012 Aug;36(8):1421-30. doi: 10.1111/j.1530-0277.2011.01716.x. Epub 2012 Feb 10. PMID 22324516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Interested candidates responded by telephone to advertisements at 5 academic centers in the United States between November 2009 and May 2010.
Pre-assignment Details: Must be alcohol dependent (DSM-IV criteria); and drinking very heavily (10 or more drinks/drinking day men; 8 or more drinks /drinking day women) 40% of the days during any consecutive 60-day interval during the 90-day period before the clinic screening visit, with at least 1 heavy drinking day occurring within the 14 days before randomization.
Groups:
- Sugar Pill and BBCET: Placebo and Brief Behavioral Compliance Enhancement Therapy
- Levetiracetam and BBCET: Levetiracetam and Brief Behavioral Therapy
Period: Overall Study
Arm/Group | Sugar Pill and BBCET | Levetiracetam and BBCET
Started | 66 | 64
Completed | 58 | 50
Not Completed | 8 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill and BBCET | Levetiracetam and BBCET | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 64 | 130
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (11.5) | 41.7 (11.7) | 44 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 52 | 47 | 99
Region of Enrollment [Number; unit: participants]
  United States | 66 | 64 | 130

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects With no Heavy Drinking Days During Study Weeks 5 Through 14.
Description: A heavy drinking day is 5+ drinks per day for men and 4+ drinks per day for women based on self report.
Time Frame: Weeks 5-14
Measure: Number; unit: percentage of subjects
Arm/Group | Sugar Pill and BBCET | Levetiracetam and BBCET
Number analyzed (Participants) | 66 | 64
percentage of subjects | 18.2 (12) | 14.1 (9)

2. Secondary Outcome: The Number of Drinks Per Drinking Day Study Weeks 5-14.
Description: based on self report
Time Frame: Study Weeks 5-14
Measure: Least Squares Mean (Standard Error); unit: drinks per day
Arm/Group | Sugar Pill and BBCET | Levetiracetam and BBCET
Number analyzed (Participants) | 66 | 64
drinks per day | 6.3 (0.58) | 7.1 (0.6)

3. Primary Outcome: The Percentage of Heavy Drinking Days Per Week During Study Weeks 5 Through 14.
Description: A heavy drinking day is 5+ drinks per day for men and 4+ drinks per day for women based on self report.
Time Frame: Study Weeks 5-14
Measure: Least Squares Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | Sugar Pill and BBCET | Levetiracetam and BBCET
Number analyzed (Participants) | 66 | 64
percentage of heavy drinking days | 41.2 (4.39) | 45.8 (4.97)

ADVERSE EVENTS:
Arm/Group | Sugar Pill and BBCET | Levetiracetam and BBCET
Serious Adverse Events (participants affected / at risk) | 10/66 | 3/64
Other Adverse Events (participants affected / at risk) | 60/66 | 58/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill and BBCET (N=66) | Levetiracetam and BBCET (N=64)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol Detoxification (Surgical and medical procedures) | 1 (1) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Clot (Vascular disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Masochism (Psychiatric disorders) | 3 (3) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill and BBCET (N=66) | Levetiracetam and BBCET (N=64)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 7 (8)
Dry Mouth (Gastrointestinal disorders) | 5 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 16 (21) | 14 (23)
Vomiting (Gastrointestinal disorders) | 8 (13) | 5 (18)
Cold Sweat (General disorders) | 1 (1) | 4 (5)
Fatigue (General disorders) | 16 (26) | 34 (47)
Irritability (General disorders) | 13 (19) | 16 (19)
Skin Laceration (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (5) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 11 (19)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7)
Agitation (Nervous system disorders) | 3 (3) | 5 (5)
Dizziness (Nervous system disorders) | 7 (8) | 8 (13)
Headache (Nervous system disorders) | 22 (47) | 22 (36)
Paraesthesia (Nervous system disorders) | 10 (13) | 5 (8)
Restlessness (Nervous system disorders) | 4 (4) | 6 (6)
Somnolence (Nervous system disorders) | 7 (8) | 10 (10)
Tremor (Nervous system disorders) | 4 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 16 (21) | 9 (12)
Depressed Mood (Psychiatric disorders) | 16 (26) | 12 (22)
Insomnia (Psychiatric disorders) | 15 (17) | 15 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 5 (6)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 10 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 8 (11)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 4 (8) | 1 (1)
Anger (Psychiatric disorders) | 3 (3) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 4 (8)
Hypertension (Vascular disorders) | 4 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No